CLINICAL TRIAL: NCT06175715
Title: The Study is Planned to Evaluate the Effectiveness and Safety of Two Types of Anesthesia (Regional and General) for Carotid Endarterectomy in 100 Patients With Acute Stage of Stroke: 50 Patients Will be Operated Under Regional Anesthesia and the Remaining 50 Patients Under General Anesthesia.
Brief Title: Regional or General Anesthesia for Carotid Endarterectomy in Patients With Acute Stage of Ischemic Stroke.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pirogov Russian National Research Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2023-11-01; First posted 2023-12-19 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Endarterectomy, Carotid

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regional anesthesia for carotid endarterectomy in patients with acute stage of ischemic stroke. (Active Comparator)
  Interventions: Procedure: carotid endarterectomy
- General anesthesia for carotid endarterectomy in patients with acute stage of ischemic stroke. (Active Comparator)
  Interventions: Procedure: carotid endarterectomy

INTERVENTIONS:
Procedure: carotid endarterectomy — carotid endarterectomy under local or general anethesia

SUMMARY:
The study is planned to evaluate the effectiveness and safety of two types of anesthesia (regional and general) for carotid endarterectomy in 100 patients with acute stage of stroke: 50 patients will be operated under regional anesthesia and the remaining 50 patients under general anesthesia.

Patient inclusion criteria:

1. Ischemic stroke in the middle cerebral artery territory
2. Ipsilateral stenosis of the internal carotid artery more than 50%
3. Neurological deficit at the time of surgical treatment: the modified Rankin scale (mRs) score of 0-4 and the US National Institutes of Health (NIHSS) stroke scale score no more than 12
4. The size of the ischemia focus: no more than 1/3 in the territory of the middle cerebral artery brain supply
5. Terms of operation: from 1 to 28 days from the moment of ischemic stroke

The primary intra-hospital and/or 30-day study endpoints:

1. Perioperative ipsilateral ischemic stroke.
2. Any stroke: contralateral ischemic or any hemorrhagic stroke.
3. Myocardial infarction.
4. Hemorrhagic complications that required surgical revision of the operating wound or transfusion of blood components.
5. Surgical site infection
6. Death
7. Main adverse cardiovascular events (stroke + myocardial infarction + death).

ELIGIBILITY:
Inclusion Criteria:

* 1. Ischemic stroke in the middle cerebral artery territory 2. Ipsilateral stenosis of the internal carotid artery more than 50% 3. Neurological deficit at the time of surgical treatment: the modified Rankin scale (mRs) score of 0-4 and the US National Institutes of Health (NIHSS) stroke scale score no more than 12 4. The size of the ischemia focus: no more than 1/3 in the territory of the middle cerebral artery brain supply 5. Terms of operation: from 1 to 28 days from the moment of ischemic stroke

Exclusion Criteria:

-

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of perioperative ipsilateral ischemic stroke (%) | in hospital, 30-day, 1 year
Rate of any stroke (%) | in hospital, 30-day, 1 year
Rate of Myocardial infarction (%) | in hospital, 30-day, 1 year
Rate of Hemorrhagic complications (%) | in hospital, 30-day, 1 year
Rate of Surgical site infection (%) | in hospital, 30-day, 1 year
Rate of Death (%) | in hospital, 30-day, 1 year
Rate of main adverse cardiovascular events (%) | in hospital, 30-day, 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Pryamikov Aleksandr, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided